CLINICAL TRIAL: NCT03279757
Title: Parameters in Fractional Laser Assisted Delivery of Topical Anesthetics: Role of Anesthetic and Application Time
Brief Title: Fractional Laser Assisted Delivery of Anesthetics IIIb
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Netherlands Institute for Pigment Disorders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NL53766.018.15b
Record Dates: First submitted 2017-09-03; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Local Anesthesia of the Skin
Keywords: Fractional laser; Topical anesthesia; Drug delivery; CO2 laser
MeSH Terms: interventions — Carticaine; Epinephrine; Lidocaine; Tetracaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- AHES 5 minutes (Experimental): This test region will be pretreated with a fractional carbon dioxide laser with a 120 μm spot at 15% density and a pulse energy of 2.5 mJ/microbeam (Fractional CO2 laser, 2.5 mJ, 15% density) in a subject blinded fashion. After pretreatment articaine hydrochloride 40 mg/ml + epinephrine 10 μg/ml solution (AHES) will be applied at this test region. 5 minutes after AHES application (under occlusion), a pain stimulus will be given at the test region with the fractional CO2 laser, 50 mJ, 5% density.
  Interventions: Drug: AHES 5 minutes; Device: fractional CO2 laser, 50 mJ, 5% density
- AHES 15 minutes (Experimental): This test region will be pretreated with a fractional carbon dioxide laser with a 120 μm spot at 15% density and a pulse energy of 2.5 mJ/microbeam (Fractional CO2 laser, 2.5 mJ, 15% density) in a subject blinded fashion. After pretreatment articaine hydrochloride 40 mg/ml + epinephrine 10 μg/ml solution (AHES) will be applied at this test region. 15 minutes after AHES application (under occlusion), a pain stimulus will be given at the test region with the fractional CO2 laser, 50 mJ, 5% density.
  Interventions: Drug: AHES 15 minutes; Device: fractional CO2 laser, 50 mJ, 5% density
- AHES 25 minutes (Experimental): This test region will be pretreated with a fractional carbon dioxide laser with a 120 μm spot at 15% density and a pulse energy of 2.5 mJ/microbeam (Fractional CO2 laser, 2.5 mJ, 15% density) in a subject blinded fashion. After pretreatment articaine hydrochloride 40 mg/ml + epinephrine 10 μg/ml solution (AHES) will be applied at this test region. 25 minutes after AHES application (under occlusion), a pain stimulus will be given at the test region with the fractional CO2 laser, 50 mJ, 5% density.
  Interventions: Drug: AHES 25 minutes; Device: fractional CO2 laser, 50 mJ, 5% density
- LTC 5 minutes (Experimental): This test region will be pretreated with a fractional carbon dioxide laser with a 120 μm spot at 15% density and a pulse energy of 2.5 mJ/microbeam (Fractional CO2 laser, 2.5 mJ, 15% density) in a subject blinded fashion. After pretreatment lidocaine 70 mg/g + tetracaine 70 mg/g cream (LTC) will be applied at this test region. 5 minutes after LTC application (under occlusion), a pain stimulus will be given at the test region with the fractional CO2 laser, 50 mJ, 5% density.
  Interventions: Drug: LTC 5 minutes; Device: fractional CO2 laser, 50 mJ, 5% density
- LTC 15 minutes (Experimental): This test region will be pretreated with a fractional carbon dioxide laser with a 120 μm spot at 15% density and a pulse energy of 2.5 mJ/microbeam (Fractional CO2 laser, 2.5 mJ, 15% density) in a subject blinded fashion. After pretreatment lidocaine 70 mg/g + tetracaine 70 mg/g cream (LTC) will be applied at this test region. 15 minutes after LTC application (under occlusion), a pain stimulus will be given at the test region with the fractional CO2 laser, 50 mJ, 5% density.
  Interventions: Drug: LTC 15 minutes; Device: fractional CO2 laser, 50 mJ, 5% density
- LTC 25 minutes (Experimental): This test region will be pretreated with a fractional carbon dioxide laser with a 120 μm spot at 15% density and a pulse energy of 2.5 mJ/microbeam (Fractional CO2 laser, 2.5 mJ, 15% density) in a subject blinded fashion. After pretreatment lidocaine 70 mg/g + tetracaine 70 mg/g cream (LTC) will be applied at this test region. 25 minutes after LTC application (under occlusion), a pain stimulus will be given at the test region with the fractional CO2 laser, 50 mJ, 5% density.
  Interventions: Drug: LTC 25 minutes; Device: fractional CO2 laser, 50 mJ, 5% density
- Unanesthetized skin (Other): A pain stimulus will be given at unanesthetized skin with the fractional CO2 laser, 50 mJ, 5% density
  Interventions: Device: fractional CO2 laser, 50 mJ, 5% density

INTERVENTIONS:
Drug: AHES 5 minutes — Topical application of AHES with 5 minutes application time After 5 minutes: pain stimulus with the fractional CO2 laser, 50 mJ, 5% density
  Other Names: Ultracain D-S forte; Articaine hydrochloride 40 mg/ml + epinephrine 10 μg/ml
  Arms: AHES 5 minutes
Drug: AHES 15 minutes — Topical application of AHES with 15 minutes application time After 15 minutes: pain stimulus with the fractional CO2 laser, 50 mJ, 5% density
  Other Names: Ultracain D-S forte; Articaine hydrochloride 40 mg/ml + epinephrine 10 μg/ml
  Arms: AHES 15 minutes
Drug: AHES 25 minutes — Topical application of AHES with 25 minutes application time After 25 minutes: pain stimulus with the fractional CO2 laser, 50 mJ, 5% density
  Other Names: Ultracain D-S forte; Articaine hydrochloride 40 mg/ml + epinephrine 10 μg/ml
  Arms: AHES 25 minutes
Drug: LTC 5 minutes — Topical application of LTC with 5 minutes application time After 5 minutes: pain stimulus with the fractional CO2 laser, 50 mJ, 5% density
  Other Names: Pliaglis cream; Lidocaine 70 mg/g + tetracaine 70 mg/g cream
  Arms: LTC 5 minutes
Drug: LTC 15 minutes — Topical application of LTC with 15 minutes application time After 15 minutes: pain stimulus with the fractional CO2 laser, 50 mJ, 5% density
  Other Names: Pliaglis cream; Lidocaine 70 mg/g + tetracaine 70 mg/g cream
  Arms: LTC 15 minutes
Drug: LTC 25 minutes — Topical application of LTC with 25 minutes application time After 25 minutes: pain stimulus with the fractional CO2 laser, 50 mJ, 5% density
  Other Names: Pliaglis cream; Lidocaine 70 mg/g + tetracaine 70 mg/g cream
  Arms: LTC 25 minutes
Device: fractional CO2 laser, 50 mJ, 5% density — Pain stimulus with the fractional CO2 laser, 50 mJ, 5% density
  Other Names: Fractional carbon dioxide laser; UltraPulse®, DeepFx handpiece; Lumenis Inc.; Ablative fractional laser

SUMMARY:
The purpose of this study are to compare the efficacy of two different commercially available local anesthetics on AFXL pretreated skin and to assess the role of the application time in this technique.

DETAILED DESCRIPTION:
Rationale: In dermatology anesthetics are frequently injected or topically applied to achieve local anesthesia. Injectable anesthetics are effective but uncomfortable during administration, especially for people who are needle phobic. Application of topical anesthesia is painless but time consuming and often only partial aesthesia is achieved due to the barrier function of the stratum corneum. (Manuskiatti, Triwongwaranat et al. 2010) Penetration of local anesthetics could be enhanced by pretreatment of the skin with ablative fractional lasers (AFXL) which locally disrupts the stratum corneum by creating an array of microscopic ablation channels. (Sklar, Burnett et al. 2014) In a previous pilot study, conducted at our institute, we demonstrated that effective anesthesia could be achieved within ten minutes after application of a topical anesthetic on skin pretreated with AFXL at painless settings. (Meesters, Bakker et al. 2015) However, little is still known about the role of the type of anesthetic the type of anesthetic and the application time on the efficacy of the anesthesia.

Objective: The objective of this study is to compare the efficacy of two different commercially available local anesthetics on AFXL pretreated skin, a low concentration articaine solution and a high concentration lidocaine/tetracaine cream. We also aim to compare the efficacy of AFXL assisted topical anesthesia after various different application times.

Study design: Prospective, single blinded, randomized, controlled, within subject, pilot study.

Study population: 15 healthy volunteers ≥18 years, who give written informed consent

Intervention: In each subject, six test regions on subject's back of 1x1 cm will be pretreated with the fractional carbon dioxide (CO2) laser at 2.5 mJ and 15% density and will be randomly allocated to application of (I) articaine hydrochloride 40 mg/ml + epinephrine 10 μg/ml 30 solution (AHES) (5 minutes application time), (II) AHES (15 minutes application time), (III) AHES (25 minutes application time), (IV) lidocaine 70 mg/g + tetracaine 70 mg/g cream (LTC) (5 minutes application time, (V) LTC (15 minutes application time), (VI) LTC (25 minutes application time). After 15 minutes a pain stimulus, consisting of a pass with the fractional CO2 laser at 50 mJ and 5% density (scanned area 6x6 mm), will be given at each test region. In addition, a reference pain stimulus with the CO2 laser at the same settings will be given at unanesthetized skin. Subjects will be asked to indicate pain on a visual analogue scale (VAS) from 0-10 (0: no pain; 10: worst imaginable pain) directly after each pain stimulus

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin type I or II
* Age ≥18 years
* Patient is willing and able to give written informed consent

Exclusion Criteria:

* History of keloid or hypertrophic scar formation or complicated wound healing
* Presence of any active skin disease
* Known allergy to local anesthesia
* Pregnancy or lactation
* Incompetency to understand what the procedure involves
* Current complaints of chronic pain or other alterations in pain sensation (e.g. due to diabetes mellitus or lepra)
* Current treatment with systemic analgesics or other medication that can influence pain sensation
* Current treatment with anticoagulants
* Fitzpatrick skin type III-VI
* Excessive sun tan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Pain score | After 5 minutes application time of the anesthetics
  The main study parameter is pain, as scored on a VAS from 0-10 (0: no pain; 10: worst imaginable pain).
Pain score | After 15 minutes application time of the anesthetics
  The main study parameter is pain, as scored on a VAS from 0-10 (0: no pain; 10: worst imaginable pain).
Pain score | After 25 minutes application time of the anesthetics
  The main study parameter is pain, as scored on a VAS from 0-10 (0: no pain; 10: worst imaginable pain).

SECONDARY OUTCOMES:
Pain score | Directly after pretreatment.
  The secondary study parameter is pain, as scored on a VAS from 0-10 (0: no pain; 10: worst imaginable pain) directly after pretreatment

CONTACTS AND LOCATIONS:
Overall Officials: Albert Wolkerstorfer, MD, PhD, Principal Investigator — Netherlands Institute for Pigment Disorders, Department of Dermatology, Academic Medical Center, University of Amsterdam; Menno A De Rie, MD, PhD, Study Director — Department of Dermatology, Academic Medical Center, University of Amsterdam

REFERENCES:
- [Background] Meesters AA, Bakker MM, de Rie MA, Wolkerstorfer A. Fractional CO2 laser assisted delivery of topical anesthetics: A randomized controlled pilot study. Lasers Surg Med. 2016 Feb;48(2):208-11. doi: 10.1002/lsm.22376. Epub 2015 May 29. PMID 26032635
- [Background] Sklar LR, Burnett CT, Waibel JS, Moy RL, Ozog DM. Laser assisted drug delivery: a review of an evolving technology. Lasers Surg Med. 2014 Apr;46(4):249-62. doi: 10.1002/lsm.22227. Epub 2014 Mar 24. PMID 24664987
- [Background] Oni G, Brown SA, Kenkel JM. Can fractional lasers enhance transdermal absorption of topical lidocaine in an in vivo animal model? Lasers Surg Med. 2012 Feb;44(2):168-74. doi: 10.1002/lsm.21130. Epub 2012 Feb 2. PMID 22302761
- [Background] Oni G, Rasko Y, Kenkel J. Topical lidocaine enhanced by laser pretreatment: a safe and effective method of analgesia for facial rejuvenation. Aesthet Surg J. 2013 Aug 1;33(6):854-61. doi: 10.1177/1090820X13496248. PMID 23908302
- [Background] Ong MW, Bashir SJ. Fractional laser resurfacing for acne scars: a review. Br J Dermatol. 2012 Jun;166(6):1160-9. doi: 10.1111/j.1365-2133.2012.10870.x. Epub 2012 May 8. PMID 22296284
- [Background] Manuskiatti W, Triwongwaranat D, Varothai S, Eimpunth S, Wanitphakdeedecha R. Efficacy and safety of a carbon-dioxide ablative fractional resurfacing device for treatment of atrophic acne scars in Asians. J Am Acad Dermatol. 2010 Aug;63(2):274-83. doi: 10.1016/j.jaad.2009.08.051. PMID 20633798
- [Background] Wolfe JW, Butterworth JF. Local anesthetic systemic toxicity: update on mechanisms and treatment. Curr Opin Anaesthesiol. 2011 Oct;24(5):561-6. doi: 10.1097/ACO.0b013e32834a9394. PMID 21841477
- [Background] Hahn IH, Hoffman RS, Nelson LS. EMLA-induced methemoglobinemia and systemic topical anesthetic toxicity. J Emerg Med. 2004 Jan;26(1):85-8. doi: 10.1016/j.jemermed.2003.03.003. PMID 14751483
- [Background] Haedersdal M, Sakamoto FH, Farinelli WA, Doukas AG, Tam J, Anderson RR. Fractional CO(2) laser-assisted drug delivery. Lasers Surg Med. 2010 Feb;42(2):113-22. doi: 10.1002/lsm.20860. PMID 20166154
- [Background] Bachhav YG, Heinrich A, Kalia YN. Controlled intra- and transdermal protein delivery using a minimally invasive Erbium:YAG fractional laser ablation technology. Eur J Pharm Biopharm. 2013 Jun;84(2):355-64. doi: 10.1016/j.ejpb.2012.11.018. Epub 2012 Nov 30. PMID 23207321
- [Background] Haak CS, Farinelli WA, Tam J, Doukas AG, Anderson RR, Haedersdal M. Fractional laser-assisted delivery of methyl aminolevulinate: Impact of laser channel depth and incubation time. Lasers Surg Med. 2012 Dec;44(10):787-95. doi: 10.1002/lsm.22102. Epub 2012 Dec 4. PMID 23212624
- [Background] Haak CS, Bhayana B, Farinelli WA, Anderson RR, Haedersdal M. The impact of treatment density and molecular weight for fractional laser-assisted drug delivery. J Control Release. 2012 Nov 10;163(3):335-41. doi: 10.1016/j.jconrel.2012.09.008. Epub 2012 Sep 21. PMID 23000695
- [Background] Tierney EP, Hanke CW. Fractionated carbon dioxide laser treatment of photoaging: prospective study in 45 patients and review of the literature. Dermatol Surg. 2011 Sep;37(9):1279-90. doi: 10.1111/j.1524-4725.2011.02082.x. PMID 22988990
- [Background] Paasch U, Haedersdal M. Laser systems for ablative fractional resurfacing. Expert Rev Med Devices. 2011 Jan;8(1):67-83. doi: 10.1586/erd.10.74. PMID 21158542
- [Background] Farkas JP, Richardson JA, Burrus CF, Hoopman JE, Brown SA, Kenkel JM. In vivo histopathologic comparison of the acute injury following treatment with five fractional ablative laser devices. Aesthet Surg J. 2010 May-Jun;30(3):457-64. doi: 10.1177/1090820X10373060. PMID 20601578
- [Background] Hantash BM, Bedi VP, Chan KF, Zachary CB. Ex vivo histological characterization of a novel ablative fractional resurfacing device. Lasers Surg Med. 2007 Feb;39(2):87-95. doi: 10.1002/lsm.20405. PMID 17115384
- [Background] Taudorf EH, Haak CS, Erlendsson AM, Philipsen PA, Anderson RR, Paasch U, Haedersdal M. Fractional ablative erbium YAG laser: histological characterization of relationships between laser settings and micropore dimensions. Lasers Surg Med. 2014 Apr;46(4):281-9. doi: 10.1002/lsm.22228. Epub 2014 Feb 5. PMID 24500855